CLINICAL TRIAL: NCT05485545
Title: Exploring Asynchronism in Operated Fallot Tetralogy : A Comparative Study of Electrical and Mechanical Activation of the Right Ventricle by Three-Dimensional Analysis
Brief Title: Asynchrony in Operated Tetralogy of Fallot
Acronym: FALLOT-XI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Reference Centre for Rare Diseases Malformations Congenital Heart Complexes (CRMR M3C-Bordeaux) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2019/39; 2021-A00770-41 (Other: ID-RCB)
Record Dates: First submitted 2022-07-26; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Tetralogy of Fallot
Keywords: FALLOT disease; CARTO; 3Dimension Echocardiography; mecanichal and electrical activation
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fallot group (Other): Patient with Fallot Tetralogy operated
  Interventions: Other: Electrophysiological exploration of the right ventricle
- Control group (Other): Patient benefiting from electrophysiological exploration for a healthy heart arrhythmia
  Interventions: Other: Electrophysiological exploration of the right ventricle

INTERVENTIONS:
Other: Electrophysiological exploration of the right ventricle — * CARTO electrophysiological mapping system
  * 3D echocardiography
  * High Resolution MRI

SUMMARY:
The objective of this work is to estimate the correlation between the electrical activation of the VD measured by the CARTO electrophysiological mapping system and the mechanical activation of the VD measured by 3D echocardiography and 3D speckle-tracking. Our hypothesis is that there is a strong correlation between electrical activation and mechanical activation in patients with an operated Fallot tetralogy.

DETAILED DESCRIPTION:
Fallot tetralogy is the most common cyanogenic congenital heart disease. Thanks to advances in surgery, most patients survive to adulthood but develop a failure of the function of the right ventricle and then of the left ventricle resulting in progressive heart failure and death of patients. Despite corrective surgeries in adulthood, including pulmonary valve surgery, heart failure remains a major problem. One of the mechanisms of this heart failure is the right intraventtricular asynchronism associated with the postoperative right branch block, which will secondaryly become complicated from an interventricular asynchronism for left intraventtricular, partly explaining the overall progressive failure of cardiac function. To date, there is no model for combining a combined analysis of electrical and mechanical activation in the same patients. Understanding these mechanisms would allow us to better understand the pathophysiology of heart failure in this population and to propose targeted therapies to prevent this asynchronism by adapting surgical techniques, or treating this asynchronism with electrical therapy such as bivascular resynchronization.

Each patient in each group will perform, according to standard practice, an electrophysiological exploration with mapping of the heart using the CARTO system, a cardiac MRI and a 3-dimensional transthoracic echocardiography.

The follow-up of each patient takes place during a scheduled hospitalization as part of the care. Their participation in the study only lasts for the duration of the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria in the Fallot group

* Male or female patient aged 18,
* Patient with Fallot Tetralogy operated.

nclusion Criteria in the Control group

* Male or female patient aged 18,
* Patient benefiting from electrophysiological exploration for a healthy heart arrhythmia,
* Patient with a significant lack of heart disease.

Exclusion Criteria:

Exclusion Criteria in the Fallot group

* Patient with associated left heart disease,
* Patient with an acoustic window that does not allow for proper echocardiography,
* Patient with contraindication to MRI,
* Woman of childbearing age without effective contraception (HAS criteria) or Pregnant (ßHCG > 20 IU/l) or nursing woman.

Exclusion Criteria in the Control group

* Patient with an acoustic window that does not allow proper echocardiography,
* Patient with MRI contraindication,
* Woman of childbearing age without effective contraception (HAS criteria) or Pregnant (ßHCG > 20 IU/l) or nursing woman,
* Cardiac pathology detected during echocardiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of electrical and mechanical activation by computational morphometry with temporal recalling to define electromechanical activation maps in healthy subjects and patients with Fallot tetralogy operated. | Day 0

SECONDARY OUTCOMES:
Area strain VD 3D global in % | Day 0
  Global 3D VD longitudinal strain in %, Global 3D VD circumferential strain in %, Mean deformation pattern, Mean RV right ventricle shape, RV Average Curvature Index.
Strain longitudinal VD 3D at the 8 segments in % | Day 0
Strain circumferential VD 3D at the 8 segments in % | Day 0
Comparison of 3D VD volume data between different populations | Day 0
  3D VD Ejection Fraction and End-Diastolic and End-Systolic Volume 3D VD; 3D right ventricle volume data processed by Tomtec 4D RV Function 2.0.
Inter-evaluator variability of 3D deformation parameters | Day 0
  Area strain 3D in %, Longitudinal strain in %, Circumferential strain in %, Global 3D at right ventricle level.
Intra-evaluator variability of 3D deformation parameters | Day 0
  Area strain 3D in %, Longitudinal strain in %, Circumferential strain in %, Global 3D at right ventricle level.
MR Analysis | Day 0
  * Right and Left Ventricular MRI Volumetry;
  * Pulmonary flow by MRI.
  * T1 spontaneous (ms) and extracellular volume fraction (%) by MRI
  * MRI scar area
Comparison of electrical activation maps based on anatomical data | Day 0
  Comparison of electrical activation maps based on anatomical data, including diffuse fibrosis and scars in Fallot subjects

CONTACTS AND LOCATIONS:
Overall Officials: Xavier IRART, MD, Study Director — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France